CLINICAL TRIAL: NCT01360515
Title: A Novel Disposable Transnasal Esophagoscope: a Prospective Pilot Trial of Feasibility, Safety and Tolerance
Brief Title: A Study of Disposable Transnasal Esophagoscope
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2010-0020
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Gastroesophageal Reflux; Esophageal Varices; Esophageal Disease
Keywords: esophagoscope; esophageal disease; gastroesophageal reflux; esophageal varices
MeSH Terms: conditions — Gastroesophageal Reflux; Esophageal and Gastric Varices; Esophageal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a pilot study of a novel disposable transnasal esophagoscope for feasibility, safety and tolerance.

DETAILED DESCRIPTION:
A disposable, transnasal esophagoscope, E.G. ScanTM was developed by IntroMedic Co. Ltd. (Seoul, Korea). This device was designed to allow patient to undergo endoscopy with minimum pain without sedation. This endoscopy system consists of thin probe with a CMOS camera, controller and simple display system. This system is light enough to carry and does occupy much space, and thus, it can be used at patient bed sides in intensive care units, in emergency rooms, and even in doctor's offices.

ELIGIBILITY:
Inclusion Criteria:

1. aged 20 years or older
2. endoscopy indicated for reflux symptoms (heartburn, epigastric soreness and/or regurgitation), dyspepsia (epigastric discomfort, bloating, early satiety), or non-cardiogenic chest pain, or known or suspected to have esophageal varices, infectious esophagitis, or other esophageal disease based on their medical history
3. a written informed consent form

Exclusion Criteria:

1. history or symptoms of severe rhinitis and sinusitis
2. symptoms of acute respiratory inflammation at the time of examination
3. abnormal anatomy of the nasal cavity or nasopharynx due to nasal tumors or previous nasopharyngeal surgery
4. taking anticoagulants such as coumadin
5. patients for whom a EGD could not be performed

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Si Young Song, M.D., Ph.D., Principal Investigator — Yonsei University
Locations (1):
- Severance Hospital, Seoul, South Korea